CLINICAL TRIAL: NCT04880148
Title: The Effectiveness of a Thyme and Honey Spray for the Management of Oral Mucositis and Xerostomia in Head and Neck Cancer Patients Undergoing Radiotherapy
Brief Title: The Effectiveness of a Thyme and Honey Spray for Oral Toxicities
Acronym: HONEY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cyprus University of Technology (Other)
Collaborators: German Oncology Center, Cyprus (Other); Bank of Cyprus Oncology Center BOCOC (Unknown)
Responsible Party: Principal Investigator, Dr. Andreas Charalambous, Associate Professor, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 21-HONEY-CUT
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Cancer of the Head and Neck; Xerostomia; Oral Mucositis; Radiation Toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Xerostomia; Stomatitis; Radiation Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thyme and Honey-based oral spray (Experimental): Thyme and Honey-based oral spray
  Interventions: Dietary Supplement: Thyme and Honey-based oral spray
- Placebo oral spray (Placebo Comparator): Placebo oral spray
  Interventions: Dietary Supplement: Placebo oral spray

INTERVENTIONS:
Dietary Supplement: Thyme and Honey-based oral spray — 4 X Sprays in the oral cavity before, immediately after and 6 hours following the radiotherapy session
  Arms: Thyme and Honey-based oral spray
Dietary Supplement: Placebo oral spray — 4 X Sprays in the oral cavity before, immediately after and 6 hours following the radiotherapy session
  Arms: Placebo oral spray

SUMMARY:
Aim: To evaluate the effectiveness of thymus honey on radiation induced-oral mucositis and xerostomia.

Background: Oral mucositis and xerostomia are two of the most severe side effects that head and neck cancer patients confront during and after the completion of radiotherapy. Although several medications are used for their treatment, these fail to provide a fully effective and comprehensive management. Honey and thyme have been studied for the management of various treatment-related side effects.

Design: Α double blinded randomised controlled trial will be used for this study.

Methods: 200 head and neck cancer patients who receive radiotherapy will be included in this study. Patients will be randomised and divided into two equal groups of 100 participants; the intervention group (oral spray with thyme and honey + standard care) and the control group ( placebo spray + standard care). Assessments with xerostomia and oral mucositis scales additionally to 4 self-administered questionnaires will occur in both groups at baseline and then weekly and 6 months following completion of treatment. The duration of the study will be 3 years from the day of approval of this research protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed histologic diagnosis of head and neck cancer
* Patients referred to non-palliative radiotherapy to the oral cavity will be included in the study
* Synchronous or induction chemotherapy, or both, will be permitted.
* Patients aged over 18,
* Patients able to provide informed consent,
* Patients having radiotherapy for at least three weeks (lower limit has been set at 50 Gy),
* Patients able to complete records accurately

Exclusion Criteria:

* Patients with a confirmed and medically treated diabetes mellitus,
* Patients with allergy to honey, thyme or any other ingredient,
* Patients who will refuse to take part in this study and
* Patients with previous radiotherapy or presence of systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Mucositis Grade (RTOG) at weekly assessments | Baseline (week 4), week 5, week 6, week 7, week 8 and week 24
  The scale includes 5 grades (from 0 to IV). Higher grade denotes more severe mucositis
Change from baseline in Xerostomia Grade (CTCAE) at weekly assessments | Baseline (week 4), week 5, week 6, week 7, week 8 and week 24
  he scale includes 5 grades (from 0 to IV). Higher grade denotes more severe xerostomia

SECONDARY OUTCOMES:
Change from baseline in Xerostomia Questionnaire (Dirix et al) | Baseline, on completion of radiotherapy, 4 weeks and 24 weeks after radiotherapy
  consists of three parts. In the first part, patients rate on a 4-likert scale (0, 1, 2, 3) the intensity of xerostomia, oral pain, taste, and dysphagia they experience and whether they suffered from more intense tooth decay or other related problems. Secondly, patients evaluate the impact of xerostomia on their Quality of Life. The Quality of Life (QoL) scales contains 15 items (ranging from 1 to 5) with a higher score indicating a worst QoL level (minimum score is 15 and the maximum is 75). Finally, patients rate the degree to which they suffered from xerostomia on a 100-mm Visual Analogue Scale (VAS).
Change from baseline in Oral Mucositis Questionnaire (OMWQ) | Baseline, on completion of radiotherapy, 4 weeks and 24 weeks after radiotherapy
  The 12-item questionnaire is designed to evaluate the overall wellbeing of the patient relating to OM during the last week. Possible answers are scored on Likert scales containing 5, 7 and 11 points. The first 2 questions assess global health and quality of life (QOL). The questions are rated on a 7-point scale, with 1 indicating very poor and 7 indicating excellent. The fourth question, which is made up of 6 items, addresses the impact of MTS on patient function and includes a 5-point scale, with 0 indicating not limited and 4 indicating unable to do. The remaining 3 questions assess the degree of mouth and throat pain and soreness using an 11-point scale, with 0 indicating no pain or soreness and 10 indicating the worst pain or soreness imaginable or possible.
Change from baseline in health-related QoL (EORTC QLQ-C30) questionnaire | Baseline, on completion of radiotherapy, 4 weeks and 24 weeks after radiotherapy
  The EORTC QLQ-C30 is a cancer-specific self-report questionnaire and comprises a global QOL scale (two items), five functional scales, three symptom scales and six single items. Scores QLQ-C30 are linearly transformed to a scale of 0-100, with a higher score indicating a better level of functioning or global QOL, or a worse level of symptoms or problems
Change from baseline in health-related QoL (EORTC QLQ-H&N43) questionnaire | Baseline, on completion of radiotherapy, 4 weeks and 24 weeks after radiotherapy
  The EORTC QLQ-H&N35 module covers specific head and neck issues, comprises ten single items and seven subscales: swallowing, senses, speech, social eating, social contact and sexuality. QLQ-H&N35 are linearly transformed to a scale of 0-100, with a higher score indicating a better level of functioning or global QOL, or a worse level of symptoms or problem.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Charalambous, PhD, Principal Investigator — Cyprus University of Technology
Locations (2):
- Cyprus (2):
  - German Oncology Center, Limassol
  - Bank of Cyprus Oncology Center, Nicosia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thrasyvoulou S, Tsitsi T, Katodritis N, Vomvas D, Charalambous M, Charalambous A. Reliability and Validity of the Greek Version of the Oral Mucositis Weekly Questionnaire in the Head and Neck Cancer Context. J Nurs Meas. 2021 Aug 1;29(2):317-333. doi: 10.1891/JNM-D-19-00096. Epub 2021 Mar 19. PMID 33741726
- [Background] Charalambous A. Hermeneutic phenomenological interpretations of patients with head and neck neoplasm experiences living with radiation-induced xerostomia: the price to pay? Eur J Oncol Nurs. 2014 Oct;18(5):512-20. doi: 10.1016/j.ejon.2014.04.007. Epub 2014 May 27. PMID 24877858
- [Result] Charalambous M, Raftopoulos V, Paikousis L, Katodritis N, Lambrinou E, Vomvas D, Georgiou M, Charalambous A. The effect of the use of thyme honey in minimizing radiation - induced oral mucositis in head and neck cancer patients: A randomized controlled trial. Eur J Oncol Nurs. 2018 Jun;34:89-97. doi: 10.1016/j.ejon.2018.04.003. Epub 2018 Apr 30. PMID 29784145
- [Result] Charalambous A, Lambrinou E, Katodritis N, Vomvas D, Raftopoulos V, Georgiou M, Paikousis L, Charalambous M. The effectiveness of thyme honey for the management of treatment-induced xerostomia in head and neck cancer patients: A feasibility randomized control trial. Eur J Oncol Nurs. 2017 Apr;27:1-8. doi: 10.1016/j.ejon.2017.01.001. Epub 2017 Jan 16. PMID 28279391